CLINICAL TRIAL: NCT06015243
Title: An Open-label, Single-arm, Multicenter, Extension Study to Evaluate the Long-term Safety and Efficacy of GR1802 Injection in Patients With Chronic Rhinosinusitis With Nasal Polyps
Brief Title: The Study of Long-term Outcomes of GR1802 in Patients With Chronic Rhinosinusitis With Nasal Polyps
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR1802-010
Record Dates: First submitted 2023-08-15; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: GR1802 (Experimental): GR1802 injection 300mg every two weeks for 16-week treatment
  Interventions: Drug: GR1802 injection

INTERVENTIONS:
Drug: GR1802 injection — 150mg/1ml. 2 ml every two weeks Route of administration: Subcutaneous

SUMMARY:
This is an open-label, single-arm, multicenter, extension study to evaluate the long-term safety and efficacy of GR1802 injection in patients with Chronic Rhinosinusitis With Nasal Polyps

DETAILED DESCRIPTION:
This trial was designed as an open, extension trial with the primary objective of evaluating the safety of long-term administration of GR1802 injection in patients with chronic rhinosinusitis with nasal polyps, and to a lesser extent, also evaluating the efficacy, immunogenicity, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Participation in a clinical study of GR1802 injection for the treatment of chronic rhinosinusitis with nasal polyps (Protocol No. GR1802-005) and fulfillment of the following: completion of prescribed treatment as required by the protocol and completion of the W16 visit.
2. the investigator judges that the subject may benefit from continued use of the test drug.
3. Able to understand and comply with the requirements of the clinical protocol, voluntarily participate in the clinical trial, and sign the informed consent form

Exclusion Criteria:

1. Poor compliance in the GR1802-005 trial and in the judgment of the investigator is unable to complete this continuation trial;
2. Use of any protocol-specified prohibited medication/treatment during the GR1802-005 trial and prior to the first dose of this study that, in the judgment of the investigator, makes continued participation in the continuation trial unsuitable.
3. The time to first dosing in the extension trial program was greater than 4 weeks from the GR1802-005 study W16 visit;
4. Nasal polyp scoring is not available for nasal polyp scores for nasal or sinus surgery (e.g., nasal polypectomy, balloon dilatation, or intranasal stent placement) that was performed prior to the first administration of the drug in the extension trial that alters the structure of the nasal sidewall;
5. Individuals who have received live/attenuated vaccination within 8 weeks prior to the first dose of the extension trial or who plan to receive live/attenuated vaccination during the trial;
6. Any serious progressive or poorly controlled concomitant disease (e.g., asthma exacerbation requiring adjustment of background medication) identified during the GR1802-005 study period for which, in the judgment of the Principal Investigator, the subject is considered unsuitable for participation in the trial;
7. Other.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-18 (Estimated); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-03-30 (Estimated)

PRIMARY OUTCOMES:
Adverse events | Baseline up to Week 24
  to characterise the safety and tolerability of GR1802 injection, including abnormal vital signs, laboratory tests, electrocardiogram.

SECONDARY OUTCOMES:
Change From Baseline at each evaluation time point in Nasal Polyp Score | Baseline up to Week 24
  NPS score ranges from 0-8. (sum of 0-4 for each nasal passage scores), higher score means a worse outcome.
Change From Baseline at each evaluation time in Nasal Congestion/Obstruction Symptom(NCS) Severity Score | Baseline up to Week 24
  Change from baseline in the NCS score. NCS score (0-3), higher score means worse nasal symptom.
Total Nasal Symptom Score(TNSS) score | Baseline up to Week 24
  Change from baseline in TNSS score. TNSS score (0-9). Higher score means worse nasal symptom.
University of Pennsylvania Smell Identification Test (UPSIT) | Baseline up to Week 24
  Change from baseline in UPSIT. UPSIT score (0-40). Higher score means better sense of smell.
Visual Analogue Scale (VAS) for Rhinosinusitis | Baseline up to Week 24
  Change from baseline in VAS score. VAS score (0-10). Higher score means worse nasal symptom.
Proportion of subjects receiving rescue therapy for nasal polyps | Baseline up to Week 24
  Rescue therapy includes Systemic Corticosteroids and endoscopic surgery
Ctrough | Baseline up to Week 24
  PK parameter: trough concentration of GR1802 injection. and exposure（CL/F, Vz/F etc.）
Vz/F | Baseline up to Week 24
  PK parameter: The volume of distribution based on the terminal elimination phase adjusted by bioavailability.
CL/F | Baseline up to Week 24
  PK parameter: The apparent volume of the central compartment cleared of drug per unit time adjusted by bioavailability.
Anti-drug antibodies(ADA) | Baseline up to Week 24
  Incidence of ADA

IPD SHARING:
Plan to Share IPD: No